CLINICAL TRIAL: NCT00003993
Title: A Phase lb Trial of the Combination of Bryostatin-1 and Low Dose Interleukin-2: Evaluation of the Functional and Molecular Status of Human Monocytes as Antigen Presenting Cells
Brief Title: Bryostatin 1 and Interleukin-2 in Treating Patients With Refractory Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067198; NCI-T99-0015; LSUMC-9901
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2006-05

CONDITIONS: Lymphoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma; unspecified adult solid tumor, protocol specific; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; primary central nervous system non-Hodgkin lymphoma; intraocular lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — aldesleukin; bryostatin 1

INTERVENTIONS:
Biological: aldesleukin
Drug: bryostatin 1

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Interleukin-2 may stimulate a person's white blood cells to kill cancer cells. Combining chemotherapy and interleukin-2 may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of interleukin-2 when given together with bryostatin 1 in treating patients with refractory solid tumors or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and side effects of bryostatin 1 and interleukin-2 in patients with refractory solid tumors or lymphomas.
* Determine the maximum tolerated dose for interleukin-2 with bryostatin 1 in these patients.
* Determine whether bryostatin 1 and interleukin-2 increase the expression of recognition and costimulatory molecules on human monocytes and their ability to act as antigen presenting cells.
* Assess any anti-tumor response in these patients treated with this regimen.

OUTLINE: This is a dose escalation study of interleukin-2.

Patients receive bryostatin 1 IV over 24 hours on days 1 and 8, and interleukin-2 subcutaneously on days 1-5 and days 8-12. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of interleukin-2 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 18-24 patients will be accrued for this study in less than 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven solid tumor or lymphoma that is not curable by surgery, radiotherapy, or standard chemotherapy, or for which no curative therapy exists
* Prostate cancer patients must have the following:

  * Tumor progression following blockade of both testicular and adrenal androgens
  * Serum testosterone in the castrate range (less than 20 ng/mL)
  * At least 3 months since prior suramin therapy
  * At least 4 weeks since prior flutamide or other antiandrogen medication and no evidence of response to treatment
  * Luprolide should continue if no prior orchiectomy
* No prior or concurrent brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0 or 1

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,500/mm^3 OR
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL

Hepatic:

* Hepatitis B surface antigen negative
* PT no greater than 14 seconds
* PTT no greater than 35 seconds
* Bilirubin no greater than 1.5 mg/dL unless due to Gilbert's disease
* SGOT and SGPT no greater than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN
* Albumin at least 2.5 g/dL

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 50 mL/min
* Corrected calcium at least 8.0 mg/dL, but no greater than 10.7 mg/dL

Cardiovascular:

* No prior myocardial infarction, coronary artery disease (CAD), congestive heart failure, second or third degree AV block, or cardiac arrhythmias requiring treatment
* No evidence of CAD on EKG

Pulmonary:

* FEV1-1 at least 70% predicted
* DLCO at least 60% predicted

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* At least 1 week since active infection requiring antibiotics
* No other medical or psychiatric condition that would preclude study
* No prior or concurrent seizure disorders controlled with medication

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior interleukin-2
* At least 4 weeks since other prior biologic therapy for solid tumors or lymphomas

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior bryostatin 1
* At least 4 weeks since other prior chemotherapy for solid tumors or lymphomas

Endocrine therapy:

* See Disease Characteristics
* At least 4 weeks since other prior endocrine therapy for solid tumors or lymphomas
* No absolute requirement for corticosteroids

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy for solid tumors or lymphomas

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior surgery for solid tumors or lymphomas

Other:

* No absolute requirement for nonsteroidal anti-inflammatory drugs or H2 blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1999-09; Primary Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Igor Espinoza-Delgado, MD, Study Chair — Gerontology Research Center
Locations (1):
- National Institute on Aging - Baltimore, Baltimore, Maryland, United States